CLINICAL TRIAL: NCT02081872
Title: Utility of PharmacoGenomics for Reducing Adverse Drug Effects
Acronym: UPGRADE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Companion Dx Reference Lab, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-101
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Genetics of Drug Metabolism
Keywords: Pharmacogenomics; Target Drug Related Adverse Events (TDAE)

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
UPGRADE aims to see whether data from Pharmacogenomic Testing (PGx) can help physicians manage patient medication regimens and assess if the testing has an effect on reducing adverse drug reactions, hospitalizations and emergency department visits.

The way an individual processes a drug is in part determined by their genes, and there is known to be genetic variation between humans in the way drugs are metabolized. The study of the way genes affect a person's response to drugs is known as "Pharmacogenomics."

ELIGIBILITY:
Inclusion Criteria:

* Subject plans to undergo current index PGx testing at the time of enrollment or underwent current index PGx testing within the prior 1-year period, for genes known to influence metabolism of at least one target drug
* Subject is aged ≥18 years
* Subject is able and willing to provide written informed consent
* Subject reveals a history of at least one TDAE or an inadequate therapeutic effect from a target drug over the 12-month period preceding expected receipt of PGx test results
* Subject is not taking an investigational medication or in an interventional trial that would interfere with participation in the registry

Exclusion Criteria:

* Subject is currently hospitalized
* Subject's medical and medication history is unavailable over the 90-day periods preceding and following the receipt of pharmacogenomic test results
* Subject is unable to provide an accurate history due to mental incapacity
* Subject is known to have undergone prior pharmacogenomic testing (exclusive of the current index PGx testing) for genes specific to the target drugs within the 2-year period preceding enrollment and these results have been previously evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects over the age of 18, receiving at least one medication with metabolism known to depend on genetic allelic variation.
Sampling Method: Non-Probability Sample
Enrollment: 279000 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Meaningful Change in Drug Regimen | 90 Days
  The primary endpoint of the study is the binary occurrence of meaningful change in drug regimen, defined for each subject as:
  * A genotype known to affect a target drug is identified by PGx testing, AND
  * The treating physician makes at least one target drug regimen change in dose, frequency, or route of administration, or when target drug discontinuation or substitutions occur.

SECONDARY OUTCOMES:
Changes in target drug regimen over the 90-day period preceding receipt of PGx results, compared to the changes made in the 90-day period thereafter | 90 days
Number of Target Drug-Related Adverse events (TDAE) over the 90-day period preceding receipt of PGx test results compared with the number over the 90-day period after the test | 90 days
Target-drug related outpatient clinic visits, emergency department visits, and hospitalizations over the 90-day period prior to the receipt of PGx test results, compared to the number of visits over the 90-day period following testing. | 90 Days

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Scottsdale Cardiovascular Center, Scottsdale, Arizona
  - ARcare, Augusta, Arkansas
  - Retina Institute of California, Arcadia, California
  - John Allen, M.D., El Cajon, California
  - Delaware Electrophysiology & Cardiology, Newark, Delaware
  - Boca Raton Clinical Research, Boca Raton, Florida
  - St. Francis Sleep, Allergy & Lung Institute, Clearwater, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Israel Machin M.D., PA, Lake Clarke Shores, Florida
  - Shaw Research Specialists, Inc., Miami, Florida
  - Angel E. Rico, M.D. PA, Miami Lakes, Florida
  - Advanced Behavioral Care, LLC, Palm Bay, Florida
  - Diverse Clinical Research Center of Chicago, LLC, Chicago, Illinois
  - Aida Mihajlovic M.D. Inc., Olympia Fields, Illinois
  - Northshore Allergy & Immunology, LLC, Covington, Louisiana
  - Centex Studies Inc, Lake Charles, Louisiana
  - B. John Hynes, M.D., Elkton, Maryland
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Pain Medicine Physicians, Millburn, New Jersey
  - Vanguard Medical Group, Montville, New Jersey
  - Virtua Medical Group, P.A., Moorestown, New Jersey
  - Coventry Cardiology Associates, Phillipsburg, New Jersey
  - Pennington Infectious Disease Associates, Trenton, New Jersey
  - White Oak Family Physicians, PA, Asheboro, North Carolina
  - Allergy Partners, P.A., Asheville, North Carolina
  - Buckeye Health and Research LLC, Hilliard, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Family Medicine and Occupational Health, Inc, Shaker Heights, Ohio
  - Lehigh Valley Hospital's Network Office of Research and innovation, Allentown, Pennsylvania
  - Wound Institute & Research Center, Dunmore, Pennsylvania
  - Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Wellmon Family Practice, Shippensburg, Pennsylvania
  - Abington Neurological Associates, LTD., Willow Grove, Pennsylvania
  - Austin, Texas
  - Harlingen, Texas
  - South Shore Medical Center, League City, Texas
  - Renaissance Psychiatry, McAllen, Texas
  - Centex Studies Inc, Pharr, Texas
  - Hillcrest Family Health Center, Waco, Texas
  - Millennium Clinical Trials LLC, Arlington, Virginia
  - Ettrick Health Center, LLC, South Chesterfield, Virginia